CLINICAL TRIAL: NCT02598375
Title: Stage 1Evaluation of Status of Early Reached Target Enteral Nutrition in Critically Ill Children in the PICU (ERTEN in PICU) Stage 2 IFABP as Biomarker of Feeding Intolerance in Critically Ill Children in the PICU(IFABP in PICU)
Brief Title: Evaluation of Status of Early Reached Target Enteral Nutrition and IFABP as Biomarker of Feeding Intolerance in Critically Ill Children
Acronym: ERTENIFABPICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Collaborators: Cukurova University (Other); Children's Medical Hospital, University of Bonn, Germany (Other); Eskisehir Osmangazi University (Other); Akdeniz University (Other); TC Erciyes University (Other); Hacettepe University (Other); Dokuz Eylul University (Other); Tepecik Training and Research Hospital (Other); Marmara University (Other); Ankara University (Other); Zonguldak Bulent Ecevit University (Other); Istanbul University (Other); Istanbul Medipol University Hospital (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other); Acibadem University (Other)
Responsible Party: Principal Investigator, Elif Keleş,MD, MD ,Resident Physician in Pediatrics, Gazi University
Other Study IDs: ERTEN-IFABP IN PICU
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Enteral Nutrition; Feeding Intolerance; Intestinal Fatty Acid Binding Protein
Keywords: Early reached target enteral nutrition in PICU feeding intolerance IFABP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples Without DNA — Urine and blood will be collected from critically ill children in PICU
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children with feeding intolerance: Critically ill children having with respiratory or catecholamine support in PICU have the feeding intolerance at least for12 hours or more.
  Interventions: Other: Feeding intolerance
- Children without feeding intolerance: Critically ill children having with respiratory or catecholamine support in PICU have not the feeding intolerance signs at least for 12 hours or less
  Interventions: Other: Feeding intolerance

INTERVENTIONS:
Other: Feeding intolerance — In this study ; it is aimed to show the value of IFABP regarding the identifying the feeding intolerance and early detection of enteral feeding intolerance

SUMMARY:
Stage 1 - Evaluation of Status of Early Reached Target Enteral Nutrition in critically ill children in the PICU (ERTEN in PICU).

In critically ill children, there is no data on the factors influenced the enteral nutrition and feeding intolerance.The investigators aim to reach these goals in our study

* To initiate the enteral feeding in pediatric intensive care units or not
* To demonstrate the reasons whether early enteral feeding is initiated or not
* To determine the incidence of feeding intolerance
* To identify the situations such as analgesia ,sedation, catecholamines or individual preferences of the medical staff which lead to delay or interruption in enteral feeding in pediatric intensive care units
* To investigate the relation between the successful enteral feeding and mortality , morbidity du to the sepsis , septic shock and multiorgan failure

Stage 2 - IFABP as biomarker of feeding intolerance in critically ill children in the PICU (IFABP in PICU)

Critically ill children are at increased risk for intestinal injury, gastrointestinal dysfunction and feeding intolerance, which are associated with delayed recovery and increased morbidity and mortality during their course in the pediatric intensive care unit. In critically ill children, there is little data on the factors influenced the enteral nutrition. We hypothesise that IFABP might be used as a biomarker which shows that the early intestinal damage due to these medications.

Aim There is no information which shows that the role of the intestinal microcirculation problems and mucosal integrity on feeding intolerance in pediatric intensive care unit.We aim to reach these goals in our study

* To show the value of IFABP regarding the identifying feeding intolerance and early detection of enteral feeding intolerance
* To show the relation between the IFABP concentration and enteral feeding intolerance
* To show the relation between the mechanical ventilation settings , sedation , inotropic medications doses and IFABP concentration and feeding intolerance
* To show the relation between IFABP concentrations and mortality and morbidity due to the sepsis , septic shock and multi system organ failure

Stage 1 (ERTEN in PICU) was completed . In many patients, initiation of feeding seems to be delayed without an evidence-based reason. ERTEN was achieved in 43 (25.3%) of 95 patients within 48 h after PICU admission. Patients with Early Initiation of Feeding were statistically significant more likely to have ERTEN. ERTEN was independent significant prognostic factors for survival (p<0.001), with reached target enteral caloric intake on day 2 indicating improved survival.

DETAILED DESCRIPTION:
Stage 1 - Evaluation of Status of Early Reached Target Enteral Nutrition in critically ill children in the PICU (ERTEN in PICU) In critically ill children, there is no data on the factors influenced the enteral nutrition and feeding intolerance.We aim to reach these goals in our study

* To initiate the enteral feeding in pediatric intensive care units or not
* To demonstrate the reasons whether early enteral feeding is initiated or not
* To determine the incidence of feeding intolerance
* To identify the situations such as analgesia ,sedation, catecholamines or individual preferences of the medical staff which lead to delay or interruption in enteral feeding in pediatric intensive care units
* To investigate the relation between the successful enteral feeding and mortality , morbidity du to the sepsis , septic shock and multiorgan failure

Stage 2 - IFABP as biomarker of feeding intolerance in critically ill children in the PICU (IFABP in PICU) Critically ill children are at increased risk for intestinal injury, gastrointestinal dysfunction and feeding intolerance, which are associated with delayed recovery and increased morbidity and mortality during their course in the pediatric intensive care unit. In critically ill children, there is little data on the factors influenced the enteral nutrition. Feeding intolerance in the critically ill children may be due to in part to alterations in gastrointestinal motility secondary to the underlying disease process or administrations of medication.It is also known the role of hyperglycemia, caloric density of enteral nutrition and gastrointestinal feedback mechanism, and routine intensive care management such as sedation, analgesia and catecholamines on the feeding intolerance in critically ill children. We hypothesise that IFABP might be used as a biomarker which shows that the early intestinal damage due to these medications.

Aim There is no information which shows that the role of the intestinal microcirculation problems and mucosal integrity on feeding intolerance in pediatric intensive care unit.We aim to reach these goals in our study

* To show the value of IFABP regarding the identifying feeding intolerance and early detection of enteral feeding intolerance
* To show the relation between the IFABP concentration and enteral feeding intolerance
* To show the relation between the mechanical ventilation settings , sedation , inotrope medications doses and IFABP concentration and feeding intolerance
* To show the relation between IFABP concentrations and mortality and morbidity due to the sepsis , septic shock and multi system organ failure We aim to reach theses goals in near future
* To find the common definitions regarding enteral feeding intolerance in order to identify and recognize the clinical problems in advance for the medical staff in Turkey
* To recognize the patients who have the possibility the enteral feeding problems with the help of the clinical and biochemical biomarkers (IFABP)
* To establish the early enteral feeding protocols in order to provide widespread using in pediatric intensive care units.
* With the help of these acquirement in the pediatrics intensive care unit to achieve the reduce the length of hospital stay , morbidity and mortality

The critically ill children who are hospitalized at least for 24 hours in PICU are eligible for the Stage 1ERTEN IN PICU

The critically ill children who are hospitalized at least for 4 days in PICU are eligible for the Stage2 IFABP IN PICU

ELIGIBILITY:
Inclusion Criteria:

* critically iil children who stayed in PICU at least for 4 days
* having informed consent from the parents of patients

Exclusion Criteria:

* children with primary gastrointestinal problems ( ulcerative colitis ,crohn ,acute gastrointestinal bleeding )

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The critically ill children in PICU who stay at least for 4 days
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
IFABP | 10 days
  IFABP level in urine will be evaluated in critically iil children in order to understand feeding intolerance and /or bacterial translocation

SECONDARY OUTCOMES:
Zonulin | 10 days
  zonulin level in blood will be evaluated in critically ill children in order to show bacterial translocation and intestinal barrier problems
8-hydroxydeoxyguanosine | 10 days
  8-hydroxydeoxyguanosine level in urine will be evaluated in critically ill children in order to show bacterial translocation and intestinal barrier problems
Claudin-3 | 10 days
  Claudin-3 level in urine will be evaluated in critically ill children in order to show bacterial translocation and intestinal barrier problems

CONTACTS AND LOCATIONS:
Overall Officials: Dincer Yildizdas, 3, Study Chair — Çukurova University Faculty of Medicine; Soyhan Bagcı, 2, Study Director — Bonn University Faculty of Medicine
Locations (1):
- Bonn University Faculty of Medicine, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is concluded the first phase of ERTEN-IFABP IN PICU.95 patients date were evaluated and the statistically significant results were obtained in the first observational phase of the study We conduct the second phase of our study.

REFERENCES:
- [Result] Mehta NM, McAleer D, Hamilton S, Naples E, Leavitt K, Mitchell P, Duggan C. Challenges to optimal enteral nutrition in a multidisciplinary pediatric intensive care unit. JPEN J Parenter Enteral Nutr. 2010 Jan-Feb;34(1):38-45. doi: 10.1177/0148607109348065. Epub 2009 Nov 10. PMID 19903872
- [Result] Lopez-Herce J. Gastrointestinal complications in critically ill patients: what differs between adults and children? Curr Opin Clin Nutr Metab Care. 2009 Mar;12(2):180-5. doi: 10.1097/MCO.0b013e3283218285. PMID 19202390
- [Result] Pathan N, Burmester M, Adamovic T, Berk M, Ng KW, Betts H, Macrae D, Waddell S, Paul-Clark M, Nuamah R, Mein C, Levin M, Montana G, Mitchell JA. Intestinal injury and endotoxemia in children undergoing surgery for congenital heart disease. Am J Respir Crit Care Med. 2011 Dec 1;184(11):1261-9. doi: 10.1164/rccm.201104-0715OC. Epub 2011 Aug 25. PMID 21868501
- [Result] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Result] Mehta NM, Compher C; A.S.P.E.N. Board of Directors. A.S.P.E.N. Clinical Guidelines: nutrition support of the critically ill child. JPEN J Parenter Enteral Nutr. 2009 May-Jun;33(3):260-76. doi: 10.1177/0148607109333114. No abstract available. PMID 19398612
- [Result] Chellis MJ, Sanders SV, Webster H, Dean JM, Jackson D. Early enteral feeding in the pediatric intensive care unit. JPEN J Parenter Enteral Nutr. 1996 Jan-Feb;20(1):71-3. doi: 10.1177/014860719602000171. PMID 8788267
- [Result] Mikhailov TA, Kuhn EM, Manzi J, Christensen M, Collins M, Brown AM, Dechert R, Scanlon MC, Wakeham MK, Goday PS. Early enteral nutrition is associated with lower mortality in critically ill children. JPEN J Parenter Enteral Nutr. 2014 May;38(4):459-66. doi: 10.1177/0148607113517903. Epub 2014 Jan 8. PMID 24403379
- [Result] Aydemir C, Dilli D, Oguz SS, Ulu HO, Uras N, Erdeve O, Dilmen U. Serum intestinal fatty acid binding protein level for early diagnosis and prediction of severity of necrotizing enterocolitis. Early Hum Dev. 2011 Oct;87(10):659-61. doi: 10.1016/j.earlhumdev.2011.05.004. Epub 2011 Jun 8. PMID 21641735
- [Result] Reisinger KW, Van der Zee DC, Brouwers HA, Kramer BW, van Heurn LW, Buurman WA, Derikx JP. Noninvasive measurement of fecal calprotectin and serum amyloid A combined with intestinal fatty acid-binding protein in necrotizing enterocolitis. J Pediatr Surg. 2012 Sep;47(9):1640-5. doi: 10.1016/j.jpedsurg.2012.02.027. PMID 22974599
- [Result] Thuijls G, van Wijck K, Grootjans J, Derikx JP, van Bijnen AA, Heineman E, Dejong CH, Buurman WA, Poeze M. Early diagnosis of intestinal ischemia using urinary and plasma fatty acid binding proteins. Ann Surg. 2011 Feb;253(2):303-8. doi: 10.1097/SLA.0b013e318207a767. PMID 21245670
- [Result] van Haren FM, Pickkers P, Foudraine N, Heemskerk S, Sleigh J, van der Hoeven JG. The effects of methylene blue infusion on gastric tonometry and intestinal fatty acid binding protein levels in septic shock patients. J Crit Care. 2010 Jun;25(2):358.e1-7. doi: 10.1016/j.jcrc.2010.02.008. Epub 2010 Apr 8. PMID 20381302
- [Result] Piton G, Belon F, Cypriani B, Regnard J, Puyraveau M, Manzon C, Navellou JC, Capellier G. Enterocyte damage in critically ill patients is associated with shock condition and 28-day mortality. Crit Care Med. 2013 Sep;41(9):2169-76. doi: 10.1097/CCM.0b013e31828c26b5. PMID 23782971